CLINICAL TRIAL: NCT06773676
Title: Evaluation of the Efficacy of a Home-Use Photobiomodulation Device for the Treatment of Patients With Knee Osteoarthritis: A Double-Blind, Randomized, Sham-Controlled Clinical Study
Brief Title: Evaluating the Effectiveness of Using a Home Laser Device to Treat Patients With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, Omri Lubovsky, Head of Orthopedic Department, Barzilai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0019-22-BRZ; MOH_2024-12-09_013784 (Registry Identifier: Israel Ministary of Health)
Record Dates: First submitted 2025-01-13; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis Of Knee
Keywords: Osteoarthritis; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Prospective, Double Blind, Randomized, Sham-Controlled, Parallel Group, Superiority comparison
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sham control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard + B-Cure Pro (Active Comparator): Subjects from the Standard + B-Cure Pro group will receive standard care and in addition will self-treat at home with the B-Cure device
  Interventions: Device: B-Cure laser pro
- Standard + Sham (Sham Comparator): Subjects from the Standard + Sham group will receive standard care and in addition will self-treat at home with the sham B-Cure device
  Interventions: Device: Sham

INTERVENTIONS:
Device: B-Cure laser pro — The B-Cure laser pro is a portal, non-invasive, photobiomodulation device, that emits light in the near infrared (808nm) over an area of 1X4.5 cm2 with power output of 250mW, and energy dose of 1J/cm2.
  Arms: Standard + B-Cure Pro
Device: Sham — The sham device is externally identical to active, emits the same guiding light and sound but does not emit the therapeutic near infrared invisible rays
  Arms: Standard + Sham

SUMMARY:
Osteoarthritis is a degenerative disease affecting joint cartilage and its surrounding tissue. It is the leading cause of disability in the elderly. Photobiomodulation (PBM), has been used widely for alleviation of pain, reduction of inflammation, and acceleration of wound healing, and particularly to treat knee osteoarthritis (KOA). The purpose of the current study is to determine if a near-infrared PBM device (B-Cure Laser), applied at home, by the patient or personal caregiver in a real-life situation, can reduce pain and improve functionality in patients with KOA.

DETAILED DESCRIPTION:
This is a prospective double blind randomized sham-controlled clinical trial. Eligible participants with KOA will be randomly allocated to receive active or sham devices for self-treatment at home in addition to standard care. Patients will be invited to the clinic for 3 visits: baseline, 1 month, and 3 months. Evaluations will include physical examination, range of motion, and patient reported outcomes including subjective pain level by visual analogue scale (VAS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), and quality of life questionnaire (SF-12). Participants will document treatments and analgesic-drug use in a diary.

The study hypothesis is that B-Cure laser treatments, applied at home by the patient, can reduce pain and improve functionality compared to standard care alone.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnoses of knee osteoarthritis by American College of Rheumatology (ACR)
2. Kellgren & Lawrence classification 1-3
3. Knee pain on movement 40 to 90 mm Visual Analog Scale
4. Knee pain and related functional reduction for at least 1 month

Exclusion Criteria:

1. Pregnant or nursing, or with the ability to become pregnant and not using an accepted form of birth control
2. Other causes of knee-related pain (e.g. hip OA, arterial insufficiency, radiculopathy etc) have been ruled out by physical examinations.
3. Knee surgery for KOA
4. Intra-articular steroid injection and/or oral steroid treatment within the last six months
5. Rheumatoid arthritis
6. Symptomatic OA in other joints (i.e. hip, hand)
7. Use of narcotics on the day of evaluation
8. Active malignancy
9. Uncontrolled diabetes mellitus
10. Neurological conditions: sciatica, neuropathy, multiple sclerosis
11. Other chronic pain conditions that may affect results: Fibromyalgia, back pain, hip pain
12. Has any photobiomodulation (low level laser) device at home or has previously used photobiomodulation for knee pain
13. Has known dermatological sensitivity to light
14. Enrolled in any other clinical trial within the last 6 weeks or enrollment in another clinical trial during participation in this trial.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-14 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in level of pain by VAS | 1month
  Subject assessment of pain will be evaluated using a Visual Analogue Scale (VAS), were 0 is "no pain" and 100 is "intolerable pain".

SECONDARY OUTCOMES:
Change from baseline in WOMAC score | 1 month
  The WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) is a disease-specific self-administered questionnaire used to assess the severity of symptoms and functional limitations in individuals with hip or knee osteoarthritis (OA). It consists of 24 items, each scored on a scale of 0-4. Higher scores indicate worse pain, stiffness, and functional limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Omri Lubovsky, MD, Principal Investigator — Barzilai University Medical Center Ashkelon Israel
Locations (1):
- Barzilai University Medical Center, Ashkelon, Southern District, Israel